CLINICAL TRIAL: NCT00386490
Title: A Phase 1, Randomized, Double-Blind, Placebo Controlled, Multi-Dose Study to Determine the Safety, Tolerance and Pharmacokinetics of 3 Dose Levels of Larazotide Acetate (AT-1001) in Healthy Volunteers
Brief Title: Safety of Larazotide Acetate in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: 9 Meters Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: CLIN1001-003
Record Dates: First submitted 2006-10-09; First posted 2006-10-11 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Healthy
Keywords: celiac disease; larazotide acetate
MeSH Terms: conditions — Celiac Disease | interventions — larazotide acetate

STUDY DESIGN:
Intervention Model Description: Phase 1, randomized, double-blind, placebo controlled multi-dose study
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Larazotide acetate 0.25 mg (Experimental): larazotide acetate 0.25 mg capsule TID for 10 days
  Interventions: Drug: larazotide acetate
- Larazotide acetate 1 mg (Experimental): larazotide acetate 1 mg capsule TID for 10 days
  Interventions: Drug: larazotide acetate
- Larazotide acetate 4 mg (Experimental): larazotide acetate 4 mg capsule TID for 10 days
  Interventions: Drug: larazotide acetate
- Placebo (Experimental): Placebo capsule TID for 10 days
  Interventions: Drug: larazotide acetate

INTERVENTIONS:
Drug: larazotide acetate — capsule for oral administration
  Other Names: AT-1001; INN-202

SUMMARY:
To demonstrate the safety, tolerance and pharmacokinetics of multiple, oral doses of larazotide acetate.

DETAILED DESCRIPTION:
CLIN1001-003 was a Phase 1, randomized, double-blind, placebo controlled multi-dose study to determine the safety, tolerance, and pharmacokinetics (including food effect) of 3 dose levels of larazotide acetate in healthy volunteers. Three (3) cohorts of 8 subjects, in which six (6) subjects in each cohort received larazotide acetate in escalating doses of 0.25 mg, 1 mg, or 4 mg TID for 10 days and two (2) subjects received placebo TID for 10 days, were studied. Subjects maintained a standard gluten-free diet. Subjects were dosed three times a day 30 minutes prior to meals except for the morning dosing on Days 1, 5, and 10. For the morning dosing on Days 1, 5, and 10 subjects, fasted overnight prior to dosing and for 2 hours post dose. Subjects were evaluated for safety (medical history, physical examination, vital signs, clinical laboratory testing, and 12-lead electrocardiograms) throughout the study. Serial blood samples were collected or pharmacokinetic determinations at baseline and 2 hours post morning dose on Days 1, 2, 5, 6 and 10.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects
* BMI between 18 and 30.

Exclusion Criteria:

* Subjects with clinically significant abnormal clinical lab results
* Hemoglobin < 12g/dL
* Subjects with diarrhea within 3 days prior to treatment visit

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2006-01-10 (Actual); Primary Completion 2006-02-27 (Actual); Study Completion 2006-02-27 (Actual)

PRIMARY OUTCOMES:
Demonstrate the safety and tolerance of multiple, oral doses of larazotide acetate | Subjects were evaluated for safety at screening, prior to administration of treatment, and following dosing of the study drug.
  Safety evaluations included medical history, physical examination, vital signs, clinical laboratory testing, and 12-lead electrocardiograms
Determine whether quantifiable concentrations of larazotide acetate are present in plasma following multiple oral doses and characterize the pharmacokinetic behavior of larazotide acetate in healthy subjects that are gluten-free and in remission | Serial blood samples were collected for pharmacokinetic determinations at baseline and 2 hours post morning dose on Days 1, 2, 5, 6 and 10.
  Pharmacokinetic samples were taken to determine whether quantifiable concentrations of larazotide acetate were present in plasma following multiple oral doses and to characterize the pharmacokinetic behavior of larazotide acetate in celiac disease subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Blake Paterson, MD, Study Chair — Alba Therapeutics
Locations (1):
- Parexel, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No